CLINICAL TRIAL: NCT05384509
Title: (COVID-19) Longitudinal Neutralizing Antibody Titers in Cancer Patients Receiving Different Anti-caner Therapies: a Retrospective Cost Research and Prospective Longitudinal Monitoring Study
Brief Title: (COVID-19) Longitudinal Neutralizing Antibody Titers in Cancer Patients Receiving Different Anti-caner Therapies
Status: Recruiting | Type: Observational
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 202101960B0
Record Dates: First submitted 2022-05-04; First posted 2022-05-20 (Actual); Last update posted 2025-02-27 (Actual); Status verified 2024-10

CONDITIONS: Cancer
Keywords: Immunotherapy; Chemotherapy; Targeted therapy; COVID-19 vaccination; Neutralizing antibody titers; Spike protein antibody titers
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Biospecimen Retention: Samples With DNA — plasma
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (4):
- Chemotherapy: Cancer Patients underwent chemotherapy
  Interventions: Diagnostic Test: solid organ malignancies treatment
- Targeted therapy: Patients underwent targeted therapy
  Interventions: Diagnostic Test: solid organ malignancies treatment
- Immunotherapy: Patients underwent immunotherapy
  Interventions: Diagnostic Test: solid organ malignancies treatment
- Disease-free: Cancer patients have been disease-free for ≥ 6 months group
  Interventions: Diagnostic Test: solid organ malignancies treatment

INTERVENTIONS:
Diagnostic Test: solid organ malignancies treatment — Major inclusion criteria for this cohort of the study included: (1) age above 20 years; (2) presence of solid organ malignancies treated with immunotherapy, chemotherapy, Target therapy irrespective of the treatment phase; and (3) eligibility for vaccination.

SUMMARY:
Patients with cancer are considered vulnerable to severe acute respiratory syndrome coronavirus 2 infection and have been prioritized in the vaccination process in several countries, including Taiwan. In addition, international oncological societies favored COVID-19 vaccination for cancer patients on the basis of risk and benefits evaluation of all available data. However, patients with cancer were excluded from severe acute respiratory syndrome coronavirus 2 vaccines registrational trials and the investigators lack data regarding the safety and efficacy of vaccination in this population. Under this perspective, the investigators undertook a large prospective study enrolling patients with solid cancers, hematologic malignancies as well as healthy volunteers for the kinetics of anti-severe acute respiratory syndrome coronavirus 2 antibodies after COVID-19 vaccination on different anticancer therapy. Major inclusion criteria for this cohort of the study included: (1) age above 20 years; (2) presence of solid organ malignancies treated with immunotherapy, chemotherapy, Targeted therapy irrespective of the treatment phase; and (3) eligibility for vaccination.

DETAILED DESCRIPTION:
Patients with cancer receiving systemic anti-cancer treatments have been generally assumed by many to be at a higher risk from the disease than their counterparts are who are not receiving anticancer treatment. However, their risk of morbidity and mortality from COVID-19 as a consequence of severe acute respiratory syndrome coronavirus 2 infection is not uniform across the world. The evidence to support this claim is scarce and limited to retrospective series arising from China, the epicenter of the COVID-19 pandemic, and involving small numbers of patients. However, despite these severe limitations, the promulgation of this hypothesis has led to widespread global changes to patterns of prescribing chemotherapy and anticancer treatment. In a global health emergency, oncologists, must secure evidence from a large datasets, which can then inform their risk-benefit analyses for individual patients in terms of the use of anticancer treatments. On March 18, 2020, the investigators launched the UK Coronavirus Cancer Monitoring Project (UKCCMP), with widespread support across our national cancer network. 8 Within 5 weeks, the UKCCMP had generated the largest prospective database of COVID-19 in patients with cancer that had been generated to date. the investigators aimed to describe the clinical and demographic characteristics and COVID-19 outcomes in this cohort of patients with cancer and symptomatic COVID-19, and attempted to assess how the presence of cancer and the receipt of cytotoxic chemotherapy and other anticancer treatments affects the COVID-19 disease phenotype.

New Taipei City Municipal Hospital has established a special infectious pneumonia ward in May 2021 to treat patients infected with symptomatic severe acute respiratory syndrome coronavirus 2 patients. During the period, 97 patients were admitted and treated with 10 infection-related deaths. In light of the current timing of the pandemic, most published serological studies are predominantly cross-sectional, or at most, include a longitudinal follow-up of few months. Severe acute respiratory syndrome coronavirus 2 has spread globally over the past year, infecting an immunologically naive population and causing significant morbidity and mortality. Immunity to severe acute respiratory syndrome coronavirus 2 induced either through natural infection or vaccination has been shown to afford a degree of protection against reinfection and/or reduce the risk of clinically significant outcomes. Seropositive recovered subjects have been estimated to have 89% protection from reinfection, and vaccine efficacies from 50 to 95% have been reported. However, the duration of protective immunity is presently unclear, primary immune responses are inevitably waning, and there is ongoing transmission of increasingly concerning viral variants that may escape control by both vaccine-induced and convalescent immune responses.

Age is considered one of the most crucial covariates that affect phenotypes. However, aging rate may vary among different populations due to genetic variation or miscellaneous environmental exposures. Chronological age is not a perfect proxy for the true biological aging status of the body. A new biological aging measure, phenotypic age (PhenoAge), has been shown to capture morbidity and mortality risk in the general US population and diverse subpopulations. However, how the phenotypic age affect host immunity is not well investigated.

There are currently no effective therapies for severe acute respiratory syndrome coronavirus 2, which causes severe respiratory illness or death. Serum neutralizing antibodies rapidly appear after severe acute respiratory syndrome coronavirus 2 infection and vaccination. However, little was known about the change of protective antibody titers both to nature infection and post vaccination. And there is ongoing transmission of increasingly concerning viral variants that may escape control by both vaccine-induced and convalescent immune responses. Defining the antibody response to severe acute respiratory syndrome coronavirus 2 in patients with cancer receiving anti-cancer therapy, (including chemotherapy, targeted therapy and immunotherapy) will be essential for understanding infection progression, long-term immunity, vaccine efficacy and how phenotypic age affect associated antibodies.

ELIGIBILITY:
Inclusion Criteria:

1. adults >20 years old;
2. cancer patients under active anti-cancer therapy, including chemotherapy (n=80), targeted therapy (n=80) and immunotherapy (n=80); and cancer patients have been disease-free for ≥ 6 months (n=80)
3. cancer patients who were full vaccinated with any brand of vaccines or cancer patients who were unvaccinated agree to complete full vaccination later.
4. patients who agreed with the content of informed consent of the study protocol.

Exclusion Criteria:

1. Patients who refused the protocol of N-antibody test and Out-Patient Departments follow-up.
2. The investigators suggest to withdraw.
3. Patient asked to withdraw from the trial at any timepoints.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: At TuCheng Hospital and Linkou Chang Gung Memorial Hospital, Cancer Patients underwent chemotherapy were enrolled as the first group (1). Patients underwent targeted therapy were enrolled as the second group (2). Cancer Patients underwent immunotherapy were enrolled as the third group (3). Cancer patients have been disease-free for ≥ 6 months group were enrolled as the fourth group (4).
Sampling Method: Probability Sample
Enrollment: 320 (Estimated)
Dates: Start 2021-12-01 (Actual); Primary Completion 2025-02-28 (Estimated); Study Completion 2025-02-28 (Estimated)

PRIMARY OUTCOMES:
COVID-19 N Ab trends among different subgroups (anti-cancer therapies) | 3 month
  COVID-19 antibodies measure after COVID-19 vaccination
COVID-19 N Ab trends among different subgroups (anti-cancer therapies) | 6 month
  COVID-19 antibodies measure after COVID-19 vaccination
COVID-19 N Ab trends among different subgroups (anti-cancer therapies) | 9 month
  COVID-19 antibodies measure after COVID-19 vaccination
COVID-19 N Ab trends among different subgroups (anti-cancer therapies) | 12 month
  COVID-19 antibodies measure after COVID-19 vaccination
COVID-19 S Ab trends among different subgroups (anti-cancer therapies) | 3 month
  COVID-19 antibodies measure after COVID-19 vaccination
COVID-19 S Ab trends among different subgroups (anti-cancer therapies) | 6 month
  COVID-19 antibodies measure after COVID-19 vaccination
COVID-19 S Ab trends among different subgroups (anti-cancer therapies) | 9 month
  COVID-19 antibodies measure after COVID-19 vaccination
COVID-19 S Ab trends among different subgroups (anti-cancer therapies) | 12 month
  COVID-19 antibodies measure after COVID-19 vaccination

SECONDARY OUTCOMES:
COVID-19 N Ab trends among different baseline PhenoAge scores | 3 month
  COVID-19 antibodies measure after COVID-19 vaccination
COVID-19 N Ab trends among different baseline PhenoAge scores | 6 month
  COVID-19 antibodies measure after COVID-19 vaccination
COVID-19 N Ab trends among different baseline PhenoAge scores | 9 month
  COVID-19 antibodies measure after COVID-19 vaccination
COVID-19 N Ab trends among different baseline PhenoAge scores | 12 month
  COVID-19 antibodies measure after COVID-19 vaccination
COVID-19 S Ab trends among different baseline PhenoAge scores | 3 month
  COVID-19 antibodies measure after COVID-19 vaccination
COVID-19 S Ab trends among different baseline PhenoAge scores | 6 month
  COVID-19 antibodies measure after COVID-19 vaccination
COVID-19 S Ab trends among different baseline PhenoAge scores | 9 month
  COVID-19 antibodies measure after COVID-19 vaccination
COVID-19 S Ab trends among different baseline PhenoAge scores | 12 month
  COVID-19 antibodies measure after COVID-19 vaccination

CONTACTS AND LOCATIONS:
Overall Officials: Chia-Hsun Hsieh, PhD, Study Director — Professor Attending Physicians
Locations (1):
- TuCheng Hospital, New Taipei City, Taiwan